CLINICAL TRIAL: NCT04584788
Title: A Single-Center, Prospective Study in Healthy Volunteers for Validation of the O3 Regional Somatic Tissue Oxygenation Monitor
Brief Title: Validation of the O3 Regional Somatic Tissue Oxygenation Monitor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCHE0001
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Results first posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-05

CONDITIONS: Oxygen Deficiency
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Healthy Adult Volunteers (Experimental): Controlled hypoxia will be induced and Masimo O3 regional oximeter-derived tissue oxygen saturation (rSO2) readings of somatic tissue will be measured. The readings will be compared with blood reference oxygen saturation values.
  Interventions: Device: Masimo O3 Regional Oximeter

INTERVENTIONS:
Device: Masimo O3 Regional Oximeter — Study sensors will be placed on somatic tissues. Readings will be taken from the tissues underneath the O3 sensors.

SUMMARY:
Testing the absolute accuracy of the Masimo O3 regional oximeter in reading somatic tissue oxygenation in healthy volunteers under controlled hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years, inclusive
* Willing and able to provide written informed consent
* Healthy subjects

Exclusion Criteria:

* Pregnant women
* Presence of any cardiovascular or pulmonary disease
* Exposure to high altitude(s) (>2000 m) within 30 days prior to the study
* Known allergy to intravenous contrast medium or heparin
* Subject has skin abnormalities affecting the digits such as psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, nail polish or acrylic nails that would prevent monitoring of SpO2 levels during the study
* Patients deemed not suitable for the study at the discretion of the Investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Site 1, Groningen, Netherlands

REFERENCES:
- [Derived] De Keijzer IN, Massari D, Niezen CK, Bokkers RPH, Vos JJ, Scheeren TWL. Agreement of somatic and renal near-infrared spectroscopy with reference blood samples during a controlled hypoxia sequence: a healthy volunteer study. J Clin Monit Comput. 2023 Jun;37(3):805-814. doi: 10.1007/s10877-022-00944-9. Epub 2022 Dec 4. PMID 36463540

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Adult Volunteers: Controlled hypoxia will be induced and Masimo O3 regional oximeter-derived rSO2 readings of somatic tissue will be measured. The readings will be compared with blood reference oxygen saturation values.
  Masimo O3 Regional Oximeter: Study sensors will be placed on somatic tissues. Readings will be taken from the tissues underneath the O3 sensors.
Period: Overall Study
Arm/Group | Healthy Adult Volunteers
Started | 37
Completed | 25
Not Completed | 12
Not completed — Physician Decision | 8
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Adult Volunteers
Number analyzed (Participants) | 25
Age, Customized [Count of Participants; unit: Participants]
  < 18 years of age | 0
  18 to 45 years of age | 25
  > 45 years of age | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of O3 Sensor by ARMS Calculation of Percent rSO2
Description: Accuracy of the sensors will be determined by comparing somatic regional oxygen saturation (rSO2) readings from the O3 sensor and blood reference oxygen saturation values and calculating the Arithmetic root mean square (ARMS).
Time Frame: 1 visit up to 8 hours
Measure: Number; unit: percentage of regional oxygen saturation
Arm/Group | Healthy Adult Volunteers
Number analyzed (Participants) | 25
percentage of regional oxygen saturation | 4.78

ADVERSE EVENTS:
Time Frame: 1 visit up to 8 hours
Arm/Group | Healthy Adult Volunteers
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 1/37
Other Adverse Events (participants affected / at risk) | 17/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Adult Volunteers (N=37)
Severe vasovagal reaction (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Adult Volunteers (N=37)
Headache (Injury, poisoning and procedural complications) | 3
Hematoma (Injury, poisoning and procedural complications) | 1
Lightheadedness (Injury, poisoning and procedural complications) | 6
Drop in blood pressure (Injury, poisoning and procedural complications) | 4
Elevated heart rate (Injury, poisoning and procedural complications) | 1
Unusual sensation near right kidney (Injury, poisoning and procedural complications) | 1
Pressure near arterial line site (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/88/NCT04584788/Prot_SAP_000.pdf